CLINICAL TRIAL: NCT01046409
Title: Comparison of Clinical, Electrical and Physiologic Significance Between Main Branch and Side Branch Vessels
Brief Title: Comparison Between Main Branch and Side Branch Vessels
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate professor, Seoul National University Hospital
Other Study IDs: H-0910-003-062
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Bifurcation; Myocardial infarction; Myocardial ischemia; Collateral
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main vessel, side branch vessel
  Interventions: Other: Measuring collateral flow

INTERVENTIONS:
Other: Measuring collateral flow — Measuring collateral flow using pressure and/or velocity coronary wire

SUMMARY:
The purpose of this trial is

1. to compare the clinical significance of the main vessel and the side branch vessel using EKG, pain score and coronary wedge pressure
2. to develop a new scoring system to predict the clinical significance of a side branch

DETAILED DESCRIPTION:
1. Clinical significance EKG change, pain score during 1 min balloon occlusion
2. Different characteristics between ST segment elevation vs non-elevation side branches
3. Comparison of coronary wedge pressure
4. Establishing a new scoring system to predict the ST elevation during 1min balloon occlusion

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Able to verbally confirm understandings of risks, benefits of receiving percutaneous coronary intervention (PCI) for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* Significant stenosis at bifurcation lesion (>50% by visual estimate) which always includes stenosis of side branch (true bifurcation)
* Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) in a native coronary artery with diameter of ≥ 2.25 mm
* Target lesion(s) amenable for PCI with final kissing balloon angioplasty for the side branch

Exclusion Criteria:

* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Patients refuse to give informed consent
* Patients with left main coronary artery stenosis
* Patients with total occlusion of the bifurcation lesion
* Patients with infarct-related artery at the lesion of interest
* Patients with left ventricular ejection fraction<40%
* Patients with primary cardiomyopathy
* Patients with chronic kidney disease defined as serum Cr>2.0
* Patients who have severe side effects or contraindication to adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant coronary artery disease, involving the bifurcation lesions
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
ST elevation during 1min balloon occlusion | Day 1 after PCI

SECONDARY OUTCOMES:
Pain score during 1min balloon occlusion | Day 1 after PCI
coronary wedge pressure | during the procedure
Usefulness of new scoring system | During the procedure
  New scoring system includes the vessel size, myocardial territory and relationship with neighboring branches

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Koo BK, Kang HJ, Youn TJ, Chae IH, Choi DJ, Kim HS, Sohn DW, Oh BH, Lee MM, Park YB, Choi YS, Tahk SJ. Physiologic assessment of jailed side branch lesions using fractional flow reserve. J Am Coll Cardiol. 2005 Aug 16;46(4):633-7. doi: 10.1016/j.jacc.2005.04.054. PMID 16098427
- [Background] Pijls NH, van Son JA, Kirkeeide RL, De Bruyne B, Gould KL. Experimental basis of determining maximum coronary, myocardial, and collateral blood flow by pressure measurements for assessing functional stenosis severity before and after percutaneous transluminal coronary angioplasty. Circulation. 1993 Apr;87(4):1354-67. doi: 10.1161/01.cir.87.4.1354. PMID 8462157
- [Background] Pijls NH, Bech GJ, el Gamal MI, Bonnier HJ, De Bruyne B, Van Gelder B, Michels HR, Koolen JJ. Quantification of recruitable coronary collateral blood flow in conscious humans and its potential to predict future ischemic events. J Am Coll Cardiol. 1995 Jun;25(7):1522-8. doi: 10.1016/0735-1097(95)00111-g. PMID 7759702
- [Background] Billinger M, Kloos P, Eberli FR, Windecker S, Meier B, Seiler C. Physiologically assessed coronary collateral flow and adverse cardiac ischemic events: a follow-up study in 403 patients with coronary artery disease. J Am Coll Cardiol. 2002 Nov 6;40(9):1545-50. doi: 10.1016/s0735-1097(02)02378-1. PMID 12427404
- [Derived] Koo BK, Lee SP, Lee JH, Park KW, Suh JW, Cho YS, Chung WY, Doh JH, Nam CW, Yu CW, Lee BK, Vassilev D, Gil R, Lim HS, Tahk SJ, Kim HS. Assessment of clinical, electrocardiographic, and physiological relevance of diagonal branch in left anterior descending coronary artery bifurcation lesions. JACC Cardiovasc Interv. 2012 Nov;5(11):1126-32. doi: 10.1016/j.jcin.2012.05.018. PMID 23174636